CLINICAL TRIAL: NCT04159649
Title: The Outcomes of ICSI Cycles With and Without Letrozole and Its Correlation With Mid-luteal Endometrial αvβ3 Integrin and Leukemia Inhibitory Factor
Brief Title: The Outcomes of ICSI Cycles With and Without Letrozole
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mansoura University (Other)
Collaborators: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Ahmed Gibreel, Assistant professor, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ZU-IRB
Record Dates: First submitted 2019-07-15; First posted 2019-11-12 (Actual); Last update posted 2019-12-16 (Actual); Status verified 2019-11

CONDITIONS: EMBRYO IMPLANTATION
MeSH Terms: interventions — Letrozole; Tablets; Gonadotropins

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- letrozole, gonadotropins and fixed GnRH antagonist (Experimental): letrozole (2.5 mg) will be given from the second day of the cycle and for 5 days, gonadotropins will be given from the third day of the cycle and GnRH antagonist will be added from the six day of the cycle for controlled ovarian stimulation in IVF (interventional group). Participant will be exposed to mid luteal endometrial sample in the pretreatment cycle. couples will be asked to use condom in the pretreatment cycle.
  Interventions: Drug: Letrozole 2.5Mg Tablet; Drug: Gonadotropins; Procedure: endometrial sample in the pretreatment cycle
- gonadotropins and fixed GnRH antagonist (control group). (Active Comparator): gonadotropins will be given from the third day of the cycle and GnRH antagonist will be added from the six day of the cycle for controlled ovarian stimulation in IVF(control group). Participant will be exposed to mid luteal endometrial sample in the pretreatment cycle. couples will be asked to use condom in the pretreatment cycle.
  Interventions: Drug: Gonadotropins; Procedure: endometrial sample in the pretreatment cycle

INTERVENTIONS:
Drug: Letrozole 2.5Mg Tablet — Gonadotropins with or letrozol in fixed Gn RH antagonist IVF protocol
  Other Names: Femara
  Arms: letrozole, gonadotropins and fixed GnRH antagonist
Drug: Gonadotropins — Gonadotropins without letrozol in fixed Gn RH antagonist IVF protocol
Procedure: endometrial sample in the pretreatment cycle — All participant will be exposed to mid luteal endometrial sample in the pretreatment cycle. couples will be asked to use condom in the pretreatment cycle.

SUMMARY:
A variety of genes working together with ovarian hormones conducts and precisely control the process of endometrial receptivity and implantation.

Leukemia inhibitory factor and αvβ3 integrin are two markers of implantation with at most importance. Reports have emphasized that these important biomarkers have a great role during the process of embryonic implantation.

αvβ3 integrin is one of the adhesion molecules which has a critical role in blastocyst apposition and attachment. Many studies have demonstrated that abnormal expression of αvβ3 integrin is associated with poor reproductive outcomes. Other studies haven't found a strong relation between αvβ3 integrin expression and reproductive outcomes Letrozole is an aromatase inhibitor which has been used in controlled ovarian stimulation especially in women with PCOS . Data suggests that letrozole addition to gonadotropins during ovarian stimulation protocols improve the response of the ovaries to FSH in low responders and increase the number of preovulatory follicles without adversely affect the outcomes.

Letrozole is used as an adjuvant therapy in ovarian stimulation protocols. So this study aims to evaluate whether the use of letrozole in combination with gonadotropins and GnRH antagonist is superior to gonadotropins and antagonist alone in women undergoing ICSI treatment.

Furthermore, both αvβ3 integrin and leukemia inhibitory factor are important markers of endometrial receptivity and implantation. Therefore, this study aims to assess the correlation between mid-luteal gene expression of both αvβ3 integrin and leukemia inhibitory factor and the clinical outcomes of antagonist cycles with or without letrozole.

DETAILED DESCRIPTION:
Embryo implantation depends on quality of the embryo, endometrial receptivity and embryo/endometrial interaction. It is estimated that two third of implantation failure is a result of defects in endometrial receptivity. A variety of genes working together with ovarian hormones conducts and precisely control the process of endometrial receptivity and implantation.

Leukemia inhibitory factor and αvβ3 integrin are two markers of implantation with at most importance. Reports have emphasized that these important bio-markers have a great role during the process of embryonic implantation . Both are expressed in the epithelial cells during the mid-secretory phase of the menstrual cycle in healthy fertile women and their absence is associated with infertility and recurrent pregnancy loss .

Leukemia inhibitory factor is a class of cytokines which plays a key role in the process of implantation in both human and animals . Studies suggest that absence of leukemia inhibitory factor in the endometrium has a negative impact on embryo implantation .

αvβ3 integrin is one of the adhesion molecules which has a critical role in blastocyst apposition and attachment. Many studies have demonstrated that abnormal expression of αvβ3 integrin is associated with poor reproductive outcomes . Other studies haven't found a strong relation between αvβ3 integrin expression and reproductive outcomes.

Letrozole is an aromatase inhibitor which has been used in controlled ovarian stimulation especially in women with PCOS . Data suggests that letrozole addition to gonadotropins during ovarian stimulation protocols improve the response of the ovaries to FSH in low responders and increase the number of preovulatory follicles without adversely affect the outcomes.

The study by Miller and his colleagues suggested that letrozole might improve αvβ3 integrin expression with possible increase in pregnancy and implantation rate. They suggested that, this drug may be a useful adjunct therapy during IVF protocols .

ELIGIBILITY:
Inclusion Criteria:

Women aged from 18 - 40 years old.

* Regular menstrual cycle (25-35).
* Women undergoing ICSI cycle

Exclusion Criteria:

Women younger than 18 or older than 40 years old.

* Women who had unilateral oophorectomy.
* Women who had uterine abnormality or pathology.
* Women who will not meet the inclusion criteria.
* Women who will refuse to participate in in the study.
* ICSI cycles with fresh or frozen TESE samples.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 224 (Estimated)
Dates: Start 2019-12-01 (Actual); Primary Completion 2020-12-30 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
ongoing pregnancy rate. | 12 weeks
  Number of pregnant women with viable fetus at 12 weeks gestation per woman randomized

SECONDARY OUTCOMES:
endometrial thickness at day of HCG administration | 9-12 days from first day of menstruation when at least three growing follicle reaches above 18 mm
  Thickness of endometrium
estrogen and progesterone levels during day of HCG, | 9-12 days from first day of menstruation when at least three growing follicle reaches above 18 mm
  estrogen and progesterone serum levels
Rate of implantation | 21 days after embryo transfer
  Number of gestational sac recognized by ultrasound in uterus 3 weeks after embryo transfer
Rate of clinical pregnancy | 5 weeks after embryo transfer
  Number of gestational sacs with evident fetal pulsations per woman randomized
miscarriage rate | 20 weeks
  Number of miscarriages per woman with positive pregnancy tests
multiple pregnancy rate | 12 weeks
  Number of multiple pregnancies per pregnant women with evident fetal pulsations
Correlation between mid-luteal gene expression of both αvβ3 integrin and leukemia inhibitory factor and the clinical outcomes of antagonist cycles with or without letrozole. | 8 weeks
  Correlation between mid-luteal gene expression of both αvβ3 integrin and leukemia inhibitory factor and the clinical outcomes of antagonist cycles with or without letrozole.

CONTACTS AND LOCATIONS:
Overall Officials: Eman ElGindy, MD, PhD, Principal Investigator — Zagazig
Locations (1):
- Mansoura University, Al Mansurah, Egypt